## CLINICAL STUDY PROTOCOL

## PROTOCOL TITLE

A DOUBLE BLIND, RANDOMIZED, PLACEBO CONTROLLED STUDY TO EVALUATE EFFICACY AND SAFETY OF "VIRACIDE" IN THE MANAGEMENT OF CORONA VIRUS DISEASE 2019 (COVID-19)

> Protocol Number: NS-VC-CT01-20 Clinicaltrial.gov ID: NCT04596085

21 Aug 2020

Confidential document Final Protocol

## STUDY SYNOPSIS

| Title | A double blind, randomized, placebo controlled study to evaluate efficacy and safety of "ViraCide" in the management of corona virus disease 2019 (COVID-19). |
|---|---|
| Study Description | This is a double blind randomized placebo controlled study will be conducted on 124 subjects, 50 years and older with mild or asymptomatic COVID-19. If symptomatic, symptoms are mild (cough, weakness, sore throat, low grade fever 38.50C, respiratory rate should not be more than 22 / min, resting SpO2 >95%, normal highly sensitive C-reactive protein (HS-CRP) (<10mg/L). There are no signs of dehydration, sepsis or shortness of breath. The study will be conducted at two centers. There will be a screening visit at Day -4 followed by three visits at the center at Days 1, 7 and 15 and a follow-up visit on Day 28. All participants will be randomized to receive either ViraCide (investigational product) or matching placebo. All subjects will receive SOC therapy. Note: If subject is discharged before Day 15 PI's discretion as per patients health condition, then assessments scheduled for Day 15 will be carried out on the discharge day (as far as possible and those not performed will be noted on appropriate CRF page) and Day 15 visit will be done telephonically. |
| Investigational<br>Product/Study drug | ViraCide softgels given per orally |
| Comparison product | Matching placebo of ViraCide softgels given per orally |
| Study Design | Double blind, randomized, placebo controlled study. Subjects will be randomized to the experimental and control groups in a 1: 1 ratio. In each group 62 subjects will be recruited, a total of 124 subjects. Subjects of the experimental arm will receive treatment with Study Drug, ViraCide and SOC. The control group will receive matching placebo and SOC. The study consists of the stages of screening, therapy, observation. There will be no switching of subjects between the arms. Participants will receive Study drug or matching placebo for 14 days during the study. |
| Sample Size | 124, including 10% dropouts |
| Study Population | <ul> <li>50 years or older</li> <li>Positive RT- PCR forSars-Co-V2.</li> <li>Either asymptomatic or have mild symptoms. Onset of symptoms within no more than 4days</li> <li>With chronic stable medical conditions: Diabetes Mellitus, or Hypertension, or chronic heart disease.</li> </ul> |
| Study Duration | Total study duration approximately 35 days Screening: 04 days Treatment duration: 14 days Follow-up: 14 days from end of treatment |

| Number of Sites | 02 (two) |
|---|---|
| Treatment Duration | 14 days |
| | , and the second |
| Treatment Arms | Two treatment arms |
| | Arm A: ViraCide softgels: 3 soft gels, two times every |
| | day after breakfast and dinner for 14 days+ SOC |
| | Therapy |
| | <ul> <li>Arm B: Placebo softgels: 3 soft gels, two times<br/>everyday after breakfast and dinner for 14 days + SOC</li> </ul> |
| | Therapy |
| Purpose of the study | To study the effectiveness and safety of the Study Drug, |
| - as possess as assaug | ViraCide |
| | softgels by oral administration compared with placebo softgels in |
| | 50 years or older subjects with asymptomatic or mildly |
| | symptomatic coronovirus infection (COVID-19) and stable |
| Objectives | comorbidities. Primary Objectives |
| Objectives | 1. To evaluate the efficacy of "ViraCide" in the management of |
| | mild COVID-19 disease |
| | Secondary Objectives |
| | 1. To evaluate the safety of "ViraCide" in the management of |
| | mild COVID-19 disease |
| Primary Endpoints | 1. TTCI using NEWS Score [Time Frame: |
| | First treatment date up to discharge day (PI's discretion as per patients health condition)] |
| | The median time in days from the start of treatment with the |
| | study drug / placebo to the persistent achievement of all of the |
| | following criteria: |
| | <ul> <li>Stopping a fever (which is defined as a decrease in</li> </ul> |
| | axillary temperature below 37 ° C without the use |
| | of anti pyretic drugs); |
| | • Respiratory rate <22 /min; |
| | <ul> <li>Oxygen saturation (SPO2) &gt; 95% when breathing<br/>in atmospheric air. Measured using pulse oximetry</li> </ul> |
| | • Systolic blood pressure ≤200mmHg |
| | <ul> <li>Pulse rate 51-90beats/minute</li> </ul> |
| | Is conscious and alert |
| | [Note: Persistent achievement means the preservation of each of |
| | the criteria for at least 7days.] |
| | 2. TTIC using 7-point ordinal scale |
| | 3. Rate of progression to severe/critical COVID-19 disease |
| | based on NEWS score [Time frame: First treatment date up to 15days] |
| | 4. Rate of progression to severe/critical COVID-19 disease |
| | based on 7-point ordinal scale [Time frame: First |
| | treatment date up to 28days] |
| | 5. Time to COVID-19 nucleic acid testing negativity in |
| | oropharyngeal/nasal swab) [Time Frame: First |
| | treatment date up to 28days] |

| Secondary Endpoints | Incidence of ICU admissions [Time Frame: 28days] |
|---|---|
| Secondary Endpoints | 2. Subject survival rate [Time Frame: 28days] |
| | 2. Subject out 11 une 11 une 2 unijoj |
| | 3. Incidence of mechanical ventilation due to COVID-19 |
| | infection [Time Frame: First treatment date up to |
| | 28days] |
| | 4. Change in clinical or laboratory assessment of comorbid |
| | condition [Time Frame: First treatment date up to |
| | 28days] |
| | 5. Percent of participants with worsening comorbid condition |
| | [Time Frame: First treatment date up to 28days] |
| | 6. Proportion of subjects in the treatment arm who |
| | had AE, SAE 7. Proportion of subjects in the placebo arm who had |
| | AE, SAE |
| Subject Selection Criteria | Inclusion criteria |
| Subject Selection Criteria | 1. 50 years or older |
| | 2. Both male and female subjects will be included |
| | 3. Positive oropharyngeal/nasal swab RT-PCR for Sars- |
| | Co- V2. Diagnosed not more than 2 days ago(diagnosis |
| | ≤2days). |
| | 4. Either asymptomatic or have mild symptoms. Onset of |
| | symptoms within no more than 4 days If symptomatic, |
| | symptoms are mild (cough, weakness, sore throat, low |
| | grade fever 38.50C, respiratory rate should not be more |
| | than 22 / min, resting SpO2 >95%, normal highly |
| | sensitive C-reactive protein (HS-CRP) (<10mg/L). There |
| | are no signs of dehydration, sepsis or shortness of |
| | breath. 5. Chronic stable medical conditions: diabetes mellitus or |
| | 5. Chronic stable medical conditions: diabetes mellitus, or hypertension, or chronic heart disease. Under treatment |
| | and controlled by medication |
| | 6. Signed informed consent/or consent given through text |
| | message, WhatsApp ore-mail. |
| | 7. Ability to understand the requirements of the Research |
| | Protocol and follow the research procedures. |
| | 8. Subject should be willing to be managed in isolation |
| | wards |
| | 9. Negative pregnancy test (for female participants) |
| | 10. Adequate contraception for study duration |
| | Exclusion criteria |
| | 1. Less than 50 years |
| | 2. With severe COVID-19 symptoms requiring immediate |
| | hospitalization |
| | 3. Investigator considers the subject unsuitable for ViraCide |
| | 4. History of symptoms of more than 4days |
| | 5. COVID-19 diagnosed >2 days ago using |
| | oropharyngeal/nasal swab RT-PCR forSars-Co- |
| | V2 6 History of cardionulmonary regugaitation |
| | 6. History of cardiopulmonary resuscitation |

| | 7. Subjects having history of organ failure or conditions |
|---|---|
| | requiring ICU monitoring and treatment, such as severe |
| | liver disease, severe renal dysfunction, upper |
| | gastrointestinal hemorrhage, disseminated intravascular |
| | coagulation or any other condition that in the PI's |
| | opinion makes the subject unfit to participate |
| | 8. Respiratory failure, ARDS or need of mechanical |
| | ventilation |
| | 9. History of acute exacerbation of comorbidity like heart |
| | failure, diabetic ketoacidosis, myocardial infection, |
| | major cardiac rhythm disorder or any other condition that |
| | in the PI"s opinion makes the subject unfit to participate |
| | 10. History of or current hepatic failure or severely |
| | compromised liver function, or renal failure or |
| | having chronic kidney disease or acute renal failure |
| | 11. History of or currently receiving treatment for an |
| | endocrine disorder like hypothyroidism, hyperthyroidism |
| | that is likely to affect the basal heart rate. |
| | 12. History of or currently under treatment for asthma |
| | [exception: patients with history of asthma, not on |
| | medications/inhalers/nebulizers for at least 6 |
| | months |
| | before study start), COPD, bronchiectasis, asbestosis and other |
| | such chronic lung conditions that can compromise SpO2 |
| | and RR. |
| | 13. HIV, HBsAg, HCV positive |
| | 14. Any condition causing immunodeficiency |
| | 15. Systemic connective tissue disease or any autoimmune |
| | disease that is likely to affect HS-CRP levels |
| | 16. History of epilepsy/epileptic fit/convulsions in last 6 |
| | months or currently on treatment for it |
| | 17. History of or currently having malignancy and |
| | being treated for it. (exception: histologically |
| | confirmed and cured carcinoma in situ) |
| | 18. Hypersensitivity reaction to Study drug/placebo |
| | 19. Any psychiatric issue for which the subject is currently |
| | undergoing treatment |
| | 20. Any history of drug/alcohol dependence within 30 |
| | days of screening or current drug/alcohol dependence |
| | 21. Inability to understand the requirements of the |
| | Research Protocol and follow the research procedures. |
| | 22. Pregnant or lactating; |
| | 23. Not willing to use adequate contraception during |
| | study duration |
| | 24. Participation in any other clinical study less than |
| | 3months before the start of the study. |
| Stopping the Study Drug | Completing 14 days of treatment |
| | 2. Progression to severe COVID-19: ViraCide will be |
| | stopped if subjects progresses to severe COVID-19 and |
| | require ICU admission, mechanical ventilation and any |
| | such situation where according to the PI the subject |

| | 17010001 |
|---|---|
| | cannot continue ViraCide. However, subject will be |
| | followed-up to capture data on ICU admission, incidence |
| | and mortality |
| | 3. Progression of comorbid condition requiring admission |
| | to ICU or inability of the subject to take anything |
| | orally. However, subject will be followed-up to capture |
| | data on ICU admission, incidence and mortality |
| | 4. Subject's participation to the study is terminated |
| | 5. Study is terminated |
| Termination of Subject's | Any participant can be removed from the study: |
| Participation in the Study | 1. By his/her own free will to not continue in the |
| | study. Subject withdrawal of informed consent. |
| | 2. Loss of contact with the subject during the study. |
| | 3. Does not comply with dosing schedule (75%-125% non- |
| | compliance) |
| | 4. The development of AE / SAE requiring the withdrawal of |
| | the study drug. However all AE / SAE will be followed-up |
| | till the study duration |
| | 5. Pregnancy confirmed anytime during the study duration |
| | 6. Another reason, which, according to the PI, requires the |
| | termination of the subject's participation in the study. |
| Study Termination | The study can be terminated if |
| | 1. There is a major deviation in Protocol |
| | 2. Another reason, which, according to the PI, |
| | requires study termination |
| Visits of Assessment | Screening and 3 visits and one telephonic follow-up |
| | Screening Lacksian (Franksian Criteria Sakinet Inform Consent |
| | Inclusion/Exclusion Criteria, Subject Inform Consent, Demography, Medical History, Physical Examination, Vital |
| | Signs, HIV; HBsAg; HCV; Hs-CRP; Pulse oximetry; |
| | NEWS scoring; 7- point ordinal scoring; Medication list |
| | review (medications being taken for comorbid conditions), |
| | Lab assessment; Urine analysis Note: Patients who do not |
| | meet the study inclusion exclusion criteria during screening |
| | should not be randomized into the study. |
| | should not be fundomized into the study. |
| | Day 1 |
| | Randomization, Vital Signs, Pulse oximetry, AE/SAE, |
| | Concomitant Medication, ViraCide/ Placebo treatment |
| | start, NEWS scoring; 7-point ordinal scoring |
| | Day 7 |
| | Physical Examination, Vital Signs, AE/SAE, Concomitant |
| | Medication, ViraCide/ Placebo Compliance check, Pulse |
| | oximetry; NEWS scoring; 7-point ordinal scoring. |
| | (Note: If the subject is discharged on this day as per PI's |
| | discretion and patient's health condition then assessment |
| | scheduled for day 15 will be carried out on discharge day). |
| | Doy 15 |
| | Day 15 Physical Examination Vital Signs, AE/SAE Concomitant |
| | Physical Examination, Vital Signs, AE/SAE, Concomitant |
| | Medication, ViraCide/ Placebo treatment end, RT-PCR for |

| | Sars- Co-V2, Hs-CRP, Safety Lab Tests, Pulse oximetry;<br>NEWS scoring; 7-point ordinal scoring, ViraCide/ Placebo<br>Compliance check, Lab assessment including urine analysis |
|---|---|
| | Day 28 Phone call follow up for time: until negative RT-PCR for Sars-Co- V2, COVID-19 related mortality, development of any COVID-19 symptom, development of any worsening of comorbid condition; Development of new AE/SAE; Resolution status of previous AE/SAEs |
| | Note: If subject is discharged before Day 15on PI's discretion as per patients health condition, then assessments scheduled for Day 15 will be carried out on the discharge day (as far as possible and those not performed will be noted on appropriate CRF page) and Day 15 visit will be done telephonically. |
| Laboratory Investigations | Screening: Recording RT-PCR- Sars-Co-V2 result; Urine pregnancy test; HIV; HBsAg; HCV;Hs-CRP; Hematology* + Biochemistry +Urine analysis*; ECG |
| | Day 1: No labs |
| | Day 7: No labs |
| | Day 15: Oropharyngeal/nasal swab for PCR- Sars-Co-V2;<br>Hematology* + Biochemistry + Urine analysis*; ECG;<br>Serological biomarker: Hs-CRP |
| | Note: *Hematology: Complete blood count (CBC); erythrocyte sedimentation rate (ESR) *Biochemistry: • Random Blood Sugar, • Serum Creatinine • SGOT,SGPT • Alkaline Phosphatase • Bilirubin-Total/Direct/Indirect • Total Proteins/Albumin/Globulin/A:Gratio • Low density lipoprotein (LDL) Cholesterol(Direct) • LDH • Total Cholesterol • Triglycerides • High Sensitive C-reactive protein(HS-CRP) • BUN (Blood Urea Nitrogen) /Urea • Serum Calcium • Serum Potassium • Uric Acid *X-ray PA view is an optional test at screening. It may be done |

| | at any other time during the study if deemed necessary by<br>the Investigator |
|---|---|
| | *Urine pregnancy test (for females only) at screening |
| | Note: If subject is discharged before Day 15 PI's discretion as per patients health condition, then assessments scheduled for Day 15 will be carried out on the discharge day (as far as possible and those not performed will be noted on appropriate CRF page) and Day 15 visit will be done telephonically. |
| Standard of Care Therapy | SOC therapy for coronavirus infection (COVID-19,SARS- |
| | CoV- 2) has not been developed yet. Treatment will be given as per the discretion of the PI or as per the guidelines issued by the GOI. GOI guidelines can be accessed here: <a href="https://www.mohfw.gov.in/">https://www.mohfw.gov.in/</a> |
| <b>Concomitant Medications</b> | 1. Medications for Diabetes Mellitus |
| Allowed by the Protocol | 2. Medications for hypertension |
| | 3. Statins |
| | 4. Blood thinners like aspirin at PI discretion |
| | 5. Any medication deemed necessary by the PI to manage the AE/SAE |
| | 6. Any other medication deemed necessary by the PI to manage a comorbid condition that is not likely to affect the treatment Protocol |
| Prohibited Concomitant<br>Medications | Any other herbal medicine or dietary supplement |
| Statistical Analysis | Sample size of total 112(56 cases in each arm) completed cases needed to assess the study objective at 80% power and 5% level of significance. Considering 10 % dropout total 124 (62 cases in each arm) |
| | cases will be enrolled in this study. |